CLINICAL TRIAL: NCT02207816
Title: Extension to Study MALARIA-055 PRI (NCT00866619) for Evaluation of Long-term Efficacy, Safety and Immunogenicity of GSK Biologicals' Candidate Malaria Vaccine (SB257049) in Infants and Children in Africa
Brief Title: An Extension to Study MALARIA-055 PRI (NCT00866619) to Evaluate the Long-term Efficacy, Safety and Immunogenicity of GSK Biologicals' Candidate Malaria Vaccine in Infants and Children in Africa
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 200599
Record Dates: First submitted 2014-07-31; First posted 2014-08-04 (Estimated); Results first posted 2019-08-15 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Malaria
Keywords: Infants; Efficacy; Children; Malaria; Plasmodium falciparum; Safety; Surveillance; Immunogenicity; RTS,S/AS01E; Africa
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Blood Specimen Collection; RTS malaria vaccine; serogroup C meningococcal conjugate vaccine; halofantrine

ARMS (3):
- GSK257049 Group (Experimental): Male or female infants (between and including 6 to 12 weeks of age)/children (between and including 5 to 17 months of age) received 3 doses of GSK257049 malaria vaccine (co-administered with Polio Sabin and Tritanrix HepB/Hib vaccines, for the infants subgroup) on a 0-1-2-month schedule, and a booster dose of GSK257049 malaria vaccine (co-administered with Polio Sabin, for the infants subgroup) at Month 20 during the primary study MALARIA-055 PRI (NCT00866619). Vaccines were administered intramuscularly: in the anterolateral left thigh (GSK257049 vaccine); left deltoid (GSK257049 booster dose); anterolateral right thigh (Tritanrix HepB/Hib vaccine); orally: Polio Sabin vaccine. No vaccination was administered during this study.
  Interventions: Procedure: Blood sampling; Biological: Malaria Vaccine 257049 (MALARIA-055 PRI); Biological: TritanrixHepB/Hib (MALARIA-055 PRI); Biological: Polio Sabin Oral Polio Vaccine (GSK) (MALARIA-055 PRI)
- GSK257049 Comparator Group (Active Comparator): Male or female infants (between and including 6 to 12 weeks of age)/children (between and including 5 to 17 months of age) received 3 doses of GSK257049 malaria vaccine (co-administered with Polio Sabin and Tritanrix HepB/Hib vaccines, for the infants subgroup) on 0-1-2-month schedule, and a booster dose of Menjugate vaccine (co-administered with Polio Sabin, for the infants subgroup) at Month 20 during the primary study MALARIA-055 PRI (NCT00866619). Vaccines were administered intramuscularly: in the anterolateral left thigh (GSK257049 vaccine); anterolateral right thigh (Tritanrix HepB/Hib vaccine); orally: Polio Sabin vaccine. No vaccination was administered during this study.
  Interventions: Procedure: Blood sampling; Biological: Malaria Vaccine 257049 (MALARIA-055 PRI); Biological: Meningococcal C Conjugate Vaccine (MALARIA-055 PRI); Biological: TritanrixHepB/Hib (MALARIA-055 PRI); Biological: Polio Sabin Oral Polio Vaccine (GSK) (MALARIA-055 PRI)
- VeroRab/Menjugate Comparator Group (Active Comparator): Male or female infants (between and including 6 to 12 weeks of age)/children (between and including 5 to 17 months of age) received 3 doses of VeroRab vaccine (children subgroup) or Menjugate vaccine (co-administered with Polio Sabin and Tritanrix HepB/Hib vaccines, for the infants subgroup) on 0-1-2-month schedule, and a booster dose of Menjugate vaccine (co-administered with Polio Sabin, for the infants subgroup) at Month 20 during the primary study MALARIA-055 PRI (NCT00866619). Vaccines were administered intramuscularly: left deltoid (VeroRab vaccine and Menjugate vaccine); anterolateral right thigh (Tritanrix HepB/Hib vaccine); orally: Polio Sabin vaccine. No vaccination was administered during this study.
  Interventions: Procedure: Blood sampling; Biological: Meningococcal C Conjugate Vaccine (MALARIA-055 PRI); Biological: Cell-culture rabies vaccine (MALARIA-055 PRI); Biological: TritanrixHepB/Hib (MALARIA-055 PRI); Biological: Polio Sabin Oral Polio Vaccine (GSK) (MALARIA-055 PRI)

INTERVENTIONS:
Procedure: Blood sampling — Annual blood sampling (Year 1, Year 2 and Year 3) during the present study.
Biological: Malaria Vaccine 257049 (MALARIA-055 PRI) — Administered intramuscularly into the left deltoid, during the MALARIA-055 study (NCT00866619).
  Arms: GSK257049 Comparator Group; GSK257049 Group
Biological: Meningococcal C Conjugate Vaccine (MALARIA-055 PRI) — Administered intramuscularly into the left deltoid, during the MALARIA-055 study (NCT00866619).
  Other Names: Menjugate
  Arms: GSK257049 Comparator Group; VeroRab/Menjugate Comparator Group
Biological: Cell-culture rabies vaccine (MALARIA-055 PRI) — Administered intramuscularly into the left deltoid, during the MALARIA-055 study (NCT00866619).
  Other Names: VeroRab
  Arms: VeroRab/Menjugate Comparator Group
Biological: TritanrixHepB/Hib (MALARIA-055 PRI) — Administered intramuscularly into the left deltoid, during the MALARIA-055 study (NCT00866619).
Biological: Polio Sabin Oral Polio Vaccine (GSK) (MALARIA-055 PRI) — Administered orally, during the MALARIA-055 study (NCT00866619).

SUMMARY:
The purpose of this study is to conduct long-term surveillance for efficacy, safety and immunogenicity of the GSK Biologicals RTS,S/AS01E candidate Plasmodium falciparum malaria vaccine in infants and children in Africa following a primary vaccination series (NCT00866619). No new subjects will be enrolled in this extension study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects' parent(s)/ Legally Acceptable Representative (LARs) who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Subjects who were enrolled and who received at least one vaccine dose in the primary study MALARIA-055 PRI NCT00866619 and who did not withdraw consent (except those who moved away from the area) during the primary study MALARIA-055 PRI NCT00866619.
* Written informed consent obtained from the parent(s)/LAR(s) of the subject.

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product or planned use during the study period.

Ages: 42 Months to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3084 (Actual)
Dates: Start 2014-09-18 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- GSK Investigational Site, Ouagadougou, Burkina Faso
- GSK Investigational Site, Kisumu, Kenya
- GSK Investigational Site, Tanga, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20045

REFERENCES:
- [Background] Tinto H, Otieno W, Gesase S, Sorgho H, Otieno L, Liheluka E, Valea I, Sing'oei V, Malabeja A, Valia D, Wangwe A, Gvozdenovic E, Guerra Mendoza Y, Jongert E, Lievens M, Roman F, Schuerman L, Lusingu J. Long-term incidence of severe malaria following RTS,S/AS01 vaccination in children and infants in Africa: an open-label 3-year extension study of a phase 3 randomised controlled trial. Lancet Infect Dis. 2019 Aug;19(8):821-832. doi: 10.1016/S1473-3099(19)30300-7. Epub 2019 Jul 9. PMID 31300331

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The randomization that was performed in the primary study NCT00866619 was kept for this extension, in which subjects from 3 sites were enrolled. Subjects remained in the same groups as the ones of the primary study.
Period: Overall Study
Arm/Group | GSK257049 Group | GSK257049 Comparator Group | VeroRab/Menjugate Comparator Group
Started | 1046 | 1010 | 1028
Completed | 995 | 924 | 961
Not Completed | 51 | 86 | 67
Not completed — Serious Adverse Event | 0 | 5 | 2
Not completed — Eligibility Criteria Not Fulfilled | 2 | 1 | 2
Not completed — Withdrawal by Subject | 4 | 9 | 7
Not completed — Migrated/Moved From Study Area | 41 | 60 | 51
Not completed — Lost to Follow-up | 3 | 9 | 1
Not completed — Other | 1 | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK257049 Group | GSK257049 Comparator Group | VeroRab/Menjugate Comparator Group | Total
Number analyzed (Participants) | 1046 | 1010 | 1028 | 3084
Age, Continuous [Mean (Standard Deviation); unit: Years] | 5.25 (0.99) | 5.23 (0.99) | 5.26 (0.97) | 5.25 (0.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 517 | 480 | 515 | 1512
  Male | 529 | 530 | 513 | 1572
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African Heritage/African American | 1046 | 1010 | 1028 | 3084

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Severe Malaria Meeting Case Definition 1
Description: Case definition 1 for severe malaria was defined as an episode of malaria with positive Plasmodium falciparum asexual parasitemia (within -1 to +3 days of admission) and with one or more marker of disease severity: Prostration, respiratory distress, Blantyre score equal to or less than (≤) 2, seizures 2 or more, hypoglycemia below (<) 2.2 millimoles per liter (mmol/L), acidosis BE ≤ -10.0 mmol/L, lactate ≥ 5.0 mmol/L or anemia < 5.0 grams per deciliter (g/dL). The incidence of severe malaria for case definition 1 is expressed as a person year rate for each group (n/T), representing the number of events (n) reported over the risk period, which was counted in days and expressed as person years at risk (T).
Time Frame: From Year 0 to Year 3 (Starting January 2014 and ending December 2016)
Population: The analysis was performed on the modified Intention-to-Treat (ITT) population, which included all subjects that consented to the trial and received at least 1 dose of the corresponding study vaccine in Malaria-055 (NCT00866619) study. The analyses on the modified ITT population were performed per treatment assignment.
Measure: Number; unit: events per person-year
Groups:
- GSK257049 [5-17M] Group: Male or female children between and including 5 to 17 months of age [5-17M], who received a 3-dose primary vaccination course of the GSK257049 malaria vaccine, according to a 0-1-2 Month schedule, followed by a booster dose of the same GSK257049 vaccine, at Month 20, in study NCT00866619 (Malaria-055). Both vaccines were administered intramuscularly into the left deltoid. No vaccination was administered during this study.
- GSK257049 Comparator [5-17M] Group: Male or female children between and including 5 to 17 months of age [5-17M], who received a 3-dose primary vaccination course of the GSK257049 malaria vaccine, according to a 0-1-2 Month schedule, followed by a booster dose of Menjugate vaccine, at Month 20, in study NCT00866619 (Malaria-055). Both vaccines were administered intramuscularly into the left deltoid. No vaccination was administered during this study.
- VeroRab Comparator [5-17M] Group: Male or female children between and including 5 to 17 months of age [5-17M], who received a 3-dose primary vaccination course of the VeroRab vaccine, according to a 0-1-2 Month schedule, followed by a booster dose of Menjugate vaccine, at Month 20, in study NCT00866619 (Malaria-055). Both vaccines were administered intramuscularly into the left deltoid. No vaccination was administered during this study.
- GSK257049 [6-12W] Group: Male or female infants between and including 6 to 12 weeks of age [6-12W], who received a 3-dose primary vaccination course of the GSK257049 malaria vaccine co-administered with Polio Sabin and Tritanrix HepB/Hib vaccines, according to a 0-1-2 Month schedule, followed by a booster dose of the GSK257049 and Polio Sabin vaccines, at Month 20, in study NCT00866619 (Malaria-055). All vaccines were administered intramuscularly in the anterolateral left thigh (GSK257049 vaccine); left deltoid (GSK257049 booster dose); anterolateral right thigh (Tritanrix HepB/Hib vaccine), except for the Polio Sabin vaccine, which was given orally. No vaccination was administered during this study.
- GSK257049 Comparator [6-12W] Group: Male or female infants between and including 6 to 12 weeks of age [6-12W], who received a 3-dose primary vaccination course of the GSK257049 malaria vaccine co-administered with Polio Sabin and Tritanrix HepB/Hib vaccines, according to a 0-1-2 Month schedule, followed by a booster dose of Menjugate and Polio Sabin vaccines, at Month 20, in study NCT00866619 (Malaria-055). All vaccines were administered intramuscularly in the anterolateral left thigh (GSK257049 vaccine); left deltoid (GSK257049 booster dose); left thigh for children under 1 year and left deltoid for children above 1 year of age (Menjugate vaccine), except for the Polio Sabin vaccine, which was given orally. No vaccination was administered during this study.
- Menjugate Comparator [6-12W] Group: Male or female infants between and including 6 to 12 weeks of age [6-12W], who received a 3-dose primary vaccination course of Menjugate vaccine co-administered with Polio Sabin and Tritanrix HepB/Hib vaccines, according to a 0-1-2 Month schedule, followed by a booster dose of Menjugate and Polio Sabin vaccines, at Month 12, in study NCT00866619 (Malaria-055). All vaccines were administered intramuscularly in the left thigh for children under 1 year and left deltoid for children above 1 year of age (Menjugate vaccine); anterolateral right thigh (Tritanrix HepB/Hib vaccine), except for the Polio Sabin vaccine, which was given orally. No vaccination was administered during this study.
Arm/Group | GSK257049 [5-17M] Group | GSK257049 Comparator [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 [6-12W] Group | GSK257049 Comparator [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 594 | 561 | 593 | 459 | 456 | 442
events per person-year | 0.001 | 0.002 | 0.002 | 0.004 | 0.003 | 0.005
Statistical Analysis 1: Comparison: GSK257049 [5-17M] Group vs VeroRab Comparator [5-17M] Group; Vaccine efficacy (VE)/ incidence comparison against all episodes of severe malaria were estimated as 1-incidence ratio (IR; total number of events/follow-up time in the GSK257049 [5-17M] Group over the total number of events/follow-up time in the VeroRab Comparator [5-17M] Group); Test type: Superiority; p = 0.2235, Negative binomial regression; Mixed model without random effect [Lievens, 2011]; Vaccine efficacy = 74.38, 95% CI 2-sided [-130 to 97.14]
Statistical Analysis 2: Comparison: GSK257049 Comparator [5-17M] Group vs VeroRab Comparator [5-17M] Group; Vaccine efficacy (VE)/ incidence comparison against all episodes of severe malaria were estimated as 1-incidence ratio (IR; total number of events/follow-up time in the GSK257049 Comparator [5-17M] Group over the total number of events/follow-up time in the VeroRab Comparator [5-17M] Group); Test type: Superiority; p = 0.8972, Negative binomial regression; Mixed model without random effect [Lievens, 2011]; Vaccine efficacy = -9.57, 95% CI 2-sided [-339 to 72.64]
Statistical Analysis 3: Comparison: GSK257049 [6-12W] Group vs Menjugate Comparator [6-12W] Group; Vaccine efficacy (VE)/ incidence comparison against all episodes of severe malaria were estimated as 1-incidence ratio (IR; total number of events/follow-up time in the GSK257049 [6-12W] Group over the total number of events/follow-up time in the Menjugate Comparator [6-12W] Group); Test type: Superiority; p = 0.5333, Negative binomial regression; Mixed model without random effect [Lievens, 2011]; Vaccine efficacy = 30.58, 95% CI 2-sided [-119 to 78.00]
Statistical Analysis 4: Comparison: GSK257049 Comparator [6-12W] Group vs Menjugate Comparator [6-12W] Group; Vaccine efficacy (VE)/ incidence comparison against all episodes of severe malaria were estimated as 1-incidence ratio (IR; total number of events/follow-up time in the GSK257049 Comparator [6-12W] Group over the total number of events/follow-up time in the Menjugate Comparator [6-12W] Group); Test type: Superiority; p = 0.3523, Negative binomial regression; Mixed model without random effect [Lievens, 2011]; Vaccine efficacy = 44.20, 95% CI 2-sided [-90.9 to 83.69]

2. Primary Outcome: Incidence of Severe Malaria Meeting Case Definition 2.
Description: Case definition 2 for severe malaria was defined as an episode of malaria with positive Plasmodium falciparum asexual parasitemia (within -1 to +3 days of admission) and with one or more marker of disease severity: Prostration, respiratory distress, Blantyre score equal to or less than (≤) 2, seizures 2 or more, hypoglycemia below (<) 2.2 millimoles per liter (mmol/L), acidosis BE ≤ -10.0 mmol/L, lactate ≥ 5.0 mmol/L or anemia < 5.0 grams per deciliter (g/dL) or SAE report including preferred terms (Malaria, Plasmodium falciparum infection or Cerebral malaria) within -1 to +3 days of admission. The incidence of severe malaria for case definition 2 is expressed as a person year rate for each group (n/T), representing the number of events (n) reported over the risk period, which was counted in days and expressed as person years at risk (T).
Time Frame: From Year 0 to Year 3 (Starting January 2014 and ending December 2016)
Population: The analysis was performed on the modified Intention-to-Treat (ITT) population, which included all subjects that consented to the trial and received at least 1 dose of the corresponding vaccine in Malaria-055 (NCT00866619) study. The analyses on the modified ITT population were performed per treatment assignment.
Measure: Number; unit: events per person-year
Arm/Group | GSK257049 [5-17M] Group | GSK257049 Comparator [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 [6-12W] Group | GSK257049 Comparator [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 594 | 561 | 593 | 459 | 456 | 442
events per person-year | 0.004 | 0.007 | 0.009 | 0.007 | 0.007 | 0.011
Statistical Analysis 1: Comparison: GSK257049 [5-17M] Group vs VeroRab Comparator [5-17M] Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0930, Negative binomial regression; Mixed model without random effect [Lievens, 2011]; Vaccine efficacy = 53.68, 95% CI 2-sided [-13.7 to 81.13]
Statistical Analysis 2: Comparison: GSK257049 Comparator [5-17M] Group vs VeroRab Comparator [5-17M] Group; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.5035, Negative binomial regression; Mixed model without random effect [Lievens, 2011]; Vaccine efficacy = 23.33, 95% CI 2-sided [-67.1 to 64.82]
Statistical Analysis 3: Comparison: GSK257049 [6-12W] Group vs Menjugate Comparator [6-12W] Group; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.3504, Negative binomial regression; Mixed model without random effect [Lievens, 2011]; Vaccine efficacy = 32.08, 95% CI 2-sided [-53.1 to 69.87]
Statistical Analysis 4: Comparison: GSK257049 Comparator [6-12W] Group vs Menjugate Comparator [6-12W] Group; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.2704, Negative binomial regression; Mixed model without random effect [Lievens, 2011]; Vaccine efficacy = 37.57, 95% CI 2-sided [-44.4 to 73.01]

3. Secondary Outcome: Incidence of Clinical Malaria Meeting Case Definition
Description: Clinical malaria was defined as an episode of malaria with positive Plasmodium falciparum asexual parasitemia, accompanied by the presence of fever (axillary temperature ≥ 37.5°C ) at the time of presentation or history of fever within 24 hours of presentation and occurring in a child who was unwell and brought for treatment to a healthcare facility. The incidence of clinical malaria for case definition 1 is expressed as a person year rate for each group (n/T), representing the number of events (n) reported over the risk period, which was counted in days and expressed as person years a t risk (T). Due to late protocol approvals and retrospective data collection the sites did not collect the data according to protocol and as such the case definition cannot be applied. For the final analysis, specific case definitions based on available data were developed.
Time Frame: From Year 0 to Year 3 (Starting January 2014 and ending December 2016)
Population: as for outcome 2
Measure: Number; unit: events per person-year
Arm/Group | GSK257049 [5-17M] Group | GSK257049 Comparator [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 [6-12W] Group | GSK257049 Comparator [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 594 | 561 | 593 | 459 | 456 | 442
events per person-year | 1.079 | 1.108 | 1.016 | 1.632 | 1.563 | 1.686
Statistical Analysis 1: Comparison: GSK257049 [5-17M] Group vs VeroRab Comparator [5-17M] Group; Vaccine efficacy (VE)/ incidence comparison against all episodes of clinical malaria were estimated as 1-incidence ratio (IR; total number of events/follow-up time in the GSK257049 [5-17M] Group over the total number of events/follow-up time in the VeroRab Comparator [5-17M] Group); Test type: Superiority; p = 0.4434, Negative binomial regression; Mixed model with over-dispersion parameter estimated from the random effect [Lievens, 2011]; Vaccine efficacy = -5.26, 95% CI 2-sided [-20.0 to 7.69]
Statistical Analysis 2: Comparison: GSK257049 Comparator [5-17M] Group vs VeroRab Comparator [5-17M] Group; Vaccine efficacy (VE)/incidence comparison against all episodes of clinical malaria were estimated as 1-incidence ratio (IR; total number of events/follow-up time in the GSK257049 Comparator [5-17M] Group over the total number of events/follow-up time in the VeroRab Comparator [5-17M] Group); Test type: Superiority; p = 0.2634, Negative binomial regression; Mixed model with over-dispersion parameter estimated from the random effect [Lievens, 2011]; Vaccine efficacy = -8.10, 95% CI 2-sided [-23.9 to 5.70]
Statistical Analysis 3: Comparison: GSK257049 [6-12W] Group vs Menjugate Comparator [6-12W] Group; Vaccine efficacy (VE)/ incidence comparison against all episodes of clinical malaria were estimated as 1-incidence ratio (IR; total number of events/follow-up time in the GSK257049 [6-12W] Group over the total number of events/follow-up time in the Menjugate Comparator [6-12W] Group); Test type: Superiority; p = 0.9278, Negative binomial regression; Mixed model with over-dispersion parameter estimated from the random effect [Lievens, 2011]; Vaccine efficacy = 0.62, 95% CI 2-sided [-13.7 to 13.13]
Statistical Analysis 4: Comparison: GSK257049 Comparator [6-12W] Group vs Menjugate Comparator [6-12W] Group; Vaccine efficacy (VE)/ incidence comparison against all episodes of clinical malaria were estimated as 1-incidence ratio (IR; total number of events/follow-up time in the GSK257049 Comparator [6-12W] Group over the total number of events/follow-up time in the Menjugate Comparator [6-12W] Group); Test type: Superiority; p = 0.4189, Negative binomial regression; Mixed model with over-dispersion parameter estimated from the random effect [Lievens, 2011]; Vaccine efficacy = 5.32, 95% CI 2-sided [-8.12 to 17.09]

4. Secondary Outcome: Number of Subjects With Malaria Hospitalization Meeting Case Definition 1.
Description: Malaria hospitalization, case definition 1, was defined as a medical hospitalization with confirmed positive Plasmodium falciparum asexual parasitemia (excludes planned admissions for medical investigation/care or elective surgery and trauma).
Time Frame: From Year 0 to Year 3 (Starting January 2014 and ending December 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 [5-17M] Group | GSK257049 Comparator [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 [6-12W] Group | GSK257049 Comparator [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 594 | 561 | 593 | 459 | 456 | 442
Participants | 7 | 11 | 14 | 10 | 10 | 13
Statistical Analysis 1: Comparison: GSK257049 [5-17M] Group vs VeroRab Comparator [5-17M] Group; Vaccine efficacy (VE) was estimated as 1-the risk ratio (RR; proportion of subjects reporting events in the GSK257049 [5-17M] Group over the proportion in VeroRab Comparator [5-17M] Group) over the entire follow-up period (from Year 0 to Year 3); Test type: Superiority; p = 0.1302, Two-sided Fisher Exact test; Vaccine efficacy = 50.10, 95% CI 2-sided [-32.2 to 82.90]
Statistical Analysis 2: Comparison: GSK257049 Comparator [5-17M] Group vs VeroRab Comparator [5-17M] Group; Vaccine efficacy (VE) was estimated as 1-the risk ratio (RR; proportion of subjects reporting events in the GSK257049 Comparator [5-17M] Group over the proportion in VeroRab Comparator [5-17M] Group) over the entire follow-up period (from Year 0 to Year 3); Test type: Superiority; p = 0.6897, Two-sided Fisher Exact test; Vaccine efficacy = 16.90, 95% CI 2-sided [-96.9 to 65.90]
Statistical Analysis 3: Comparison: GSK257049 [6-12W] Group vs Menjugate Comparator [6-12W] Group; Vaccine efficacy (VE) was estimated as 1-the risk ratio (RR; proportion of subjects reporting events in the GSK257049 [6-12W] Group over the proportion in Menjugate Comparator [6-12W] Group) over the entire follow-up period (from Year 0 to Year 3); Test type: Superiority; p = 0.5299, Two-sided Fisher Exact test; Vaccine efficacy = 25.90, 95% CI 2-sided [-82.9 to 70.90]
Statistical Analysis 4: Comparison: GSK257049 Comparator [6-12W] Group vs Menjugate Comparator [6-12W] Group; Vaccine efficacy (VE) was estimated as 1-the risk ratio (RR; proportion of subjects reporting events in the GSK257049 Comparator [6-12W] Group over the proportion in Menjugate Comparator [6-12W] Group) over the entire follow-up period (from Year 0 to Year 3); Test type: Superiority; p = 0.5307, Two-sided Fisher Exact test; Vaccine efficacy = 25.40, 95% CI 2-sided [-84.1 to 70.70]

5. Secondary Outcome: Number of Subjects With Malaria Hospitalization Meeting Case Definition 2.
Description: Malaria hospitalization, case definition 2, was defined as a hospitalization for which, in the judgment of the principal investigator, Plasmodium falciparum infection was the sole or a major contributing factor to the presentation.
Time Frame: From Year 0 to Year 3 (Starting January 2014 and ending December 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 [5-17M] Group | GSK257049 Comparator [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 [6-12W] Group | GSK257049 Comparator [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 594 | 561 | 593 | 459 | 456 | 442
Participants | 7 | 8 | 13 | 10 | 9 | 14
Statistical Analysis 1: Comparison: GSK257049 [5-17M] Group vs VeroRab Comparator [5-17M] Group; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.1853, Two-sided Fisher Exact test; Vaccine efficacy = 46.20, 95% CI 2-sided [-45.0 to 81.80]
Statistical Analysis 2: Comparison: GSK257049 Comparator [5-17M] Group vs VeroRab Comparator [5-17M] Group; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p = 0.3828, Two-sided Fisher Exact test; Vaccine efficacy = 35.00, 95% CI 2-sided [-69.3 to 76.60]
Statistical Analysis 3: Comparison: GSK257049 [6-12W] Group vs Menjugate Comparator [6-12W] Group; [analysis description as in outcome 4, analysis 3]; Test type: Superiority; p = 0.4112, Two-sided Fisher Exact test; Vaccine efficacy = 31.20, 95% CI 2-sided [-66.5 to 72.70]
Statistical Analysis 4: Comparison: GSK257049 Comparator [6-12W] Group vs Menjugate Comparator [6-12W] Group; [analysis description as in outcome 4, analysis 4]; Test type: Superiority; p = 0.4121, Two-sided Fisher Exact test; Vaccine efficacy = 30.80, 95% CI 2-sided [-67.6 to 72.50]

6. Secondary Outcome: Number of Subjects With Prevalent Parasitemia
Description: Prevalent parasitemia (PP) was defined as a documented Plasmodium falciparum asexual parasite density greater than (>) 0 parasites/µL, identified at an annual visit.
Time Frame: At Years 1, 2 and 3
Population: The analysis was performed on the modified ITT population, which included all subjects that consented to the trial and received at least 1 dose of the corresponding vaccine in Malaria-055 (NCT00866619) study, with available results at the specified time-points. The analyses on the modified ITT population were performed per treatment assignment
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 [5-17M] Group | GSK257049 Comparator [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 [6-12W] Group | GSK257049 Comparator [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 565 | 525 | 561 | 436 | 435 | 420
Participants
  Prevalent parasitemia, Year 1: number analyzed (Participants) | 152 | 139 | 154 | 168 | 176 | 169
  Prevalent parasitemia, Year 1 | 52 | 46 | 89 | 48 | 65 | 61
  Prevalent parasitemia, Year 2 | 132 | 127 | 156 | 116 | 133 | 123
  Prevalent parasitemia, Year 3: number analyzed (Participants) | 561 | 515 | 549 | 434 | 408 | 411
  Prevalent parasitemia, Year 3 | 135 | 148 | 158 | 106 | 105 | 99
Statistical Analysis 1: Comparison: GSK257049 [5-17M] Group vs VeroRab Comparator [5-17M] Group; Vaccine efficacy (VE) against prevalent parasitemia assessed at Year 1 was estimated as 1-RR, where RR is the risk ratio (proportion of subjects reporting events in the GSK257049 [5-17M] Group over the proportion in VeroRab Comparator [5-17M] Group); Test type: Superiority; p < 0.0001, Two-sided Fisher Exact test; Vaccine efficacy = 40.80, 95% CI 2-sided [15.70 to 58.80]
Statistical Analysis 2: Comparison: GSK257049 Comparator [5-17M] Group vs VeroRab Comparator [5-17M] Group; Vaccine efficacy (VE) against prevalent parasitemia assessed at Year 1 was estimated as 1-RR, where RR is the risk ratio (proportion of subjects reporting events in the GSK257049 Comparator [5-17M] Group over the proportion in VeroRab Comparator [5-17M] Group); Test type: Superiority; p < 0.0001, Two-sided Fisher Exact test; Vaccine effiicacy = 42.70, 95% CI 2-sided [17.40 to 60.80]
Statistical Analysis 3: Comparison: GSK257049 [5-17M] Group vs VeroRab Comparator [5-17M] Group; Vaccine efficacy (VE) against prevalent parasitemia assessed at Year 2 was estimated as 1-RR, where RR is the risk ratio (proportion of subjects reporting events in the GSK257049 [5-17M] Group over the proportion in VeroRab Comparator [5-17M] Group); Test type: Superiority; p = 0.0883, Two-sided Fisher Exact test; Vaccine efficacy = 16.00, 95% CI 2-sided [-6.60 to 33.90]
Statistical Analysis 4: Comparison: GSK257049 Comparator [5-17M] Group vs VeroRab Comparator [5-17M] Group; Vaccine efficacy (VE) against prevalent parasitemia assessed at Year 2 was estimated as 1-RR, where RR is the risk ratio (proportion of subjects reporting events in the GSK257049 Comparator [5-17M] Group over the proportion in VeroRab Comparator [5-17M] Group); Test type: Superiority; p = 0.1889, Two-sided Fisher Exact test; Vaccine efficacy = 13.00, 95% CI 2-sided [-10.7 to 31.70]
Statistical Analysis 5: Comparison: GSK257049 [5-17M] Group vs VeroRab Comparator [5-17M] Group; Vaccine efficacy (VE) against prevalent parasitemia assessed at Year 3 was estimated as 1-RR, where RR is the risk ratio (proportion of subjects reporting events in the GSK257049 [5-17M] Group over the proportion in VeroRab Comparator [5-17M] Group); Test type: Superiority; p = 0.0770, Two-sided Fisher Exact test; Vaccine efficacy = 16.40, 95% CI 2-sided [-5.90 to 34.00]
Statistical Analysis 6: Comparison: GSK257049 Comparator [5-17M] Group vs VeroRab Comparator [5-17M] Group; Vaccine efficacy (VE) against prevalent parasitemia assessed at Year 3 was estimated as 1-RR, where RR is the risk ratio (proportion of subjects reporting events in the GSK257049 Comparator [5-17M] Group over the proportion in VeroRab Comparator [5-17M] Group); Test type: Superiority; p = 1.0000, Two-sided Fisher Exact test; Vaccine efficacy = 0.10, 95% CI 2-sided [-25.8 to 20.70]
Statistical Analysis 7: Comparison: GSK257049 [6-12W] Group vs Menjugate Comparator [6-12W] Group; Vaccine efficacy (VE) against prevalent parasitemia assessed at Year 1 was estimated as 1-RR, where RR is the risk ratio (proportion of subjects reporting events in the GSK257049 [6-12W] Group over the proportion in Menjugate Comparator [6-12W] Group); Test type: Superiority; p = 0.1624, Two-sided Fisher Exact test; Vaccine efficacy = 20.80, 95% CI 2-sided [-17.5 to 46.90]
Statistical Analysis 8: Comparison: GSK257049 Comparator [6-12W] Group vs Menjugate Comparator [6-12W] Group; Vaccine efficacy (VE) against prevalent parasitemia assessed at Year 1 was estimated as 1-RR, where RR is the risk ratio (proportion of subjects reporting events in the GSK257049 Comparator [6-12W] Group over the proportion in Menjugate Comparator [6-12W] Group); Test type: Superiority; p = 0.9112, Two-sided Fisher Exact test; Vaccine efficacy = -2.30, 95% CI 2-sided [-47.6 to 29.00]
Statistical Analysis 9: Comparison: GSK257049 [6-12W] Group vs Menjugate Comparator [6-12W] Group; Vaccine efficacy (VE) against prevalent parasitemia assessed at Year 2 was estimated as 1-RR, where RR is the risk ratio (proportion of subjects reporting events in the GSK257049 [6-12W] Group over the proportion in Menjugate Comparator [6-12W] Group); Test type: Superiority; p = 0.4023, Two-sided Fisher Exact test; Vaccine efficacy = 9.20, 95% CI 2-sided [-18.0 to 30.10]
Statistical Analysis 10: Comparison: GSK257049 Comparator [6-12W] Group vs Menjugate Comparator [6-12W] Group; Vaccine efficacy (VE) against prevalent parasitemia assessed at Year 2 was estimated as 1-RR, where RR is the risk ratio (proportion of subjects reporting events in the GSK257049 Comparator [6-12W] Group over the proportion in Menjugate Comparator [6-12W] Group); Test type: Superiority; p = 0.7091, Two-sided Fisher Exact test; Vaccine efficacy = -4.40, 95% CI 2-sided [-34.5 to 18.90]
Statistical Analysis 11: Comparison: GSK257049 [6-12W] Group vs Menjugate Comparator [6-12W] Group; Vaccine efficacy (VE) against prevalent parasitemia assessed at Year 3 was estimated as 1-RR, where RR is the risk ratio (proportion of subjects reporting events in the GSK257049 [6-12W] Group over the proportion in Menjugate Comparator [6-12W] Group); Test type: Superiority; p = 0.9361, Two-sided Fisher Exact test; Vaccine efficacy = -1.40, 95% CI 2-sided [-34.7 to 23.60]
Statistical Analysis 12: Comparison: GSK257049 Comparator [6-12W] Group vs Menjugate Comparator [6-12W] Group; Vaccine efficacy (VE) against prevalent parasitemia assessed at Year 3 was estimated as 1-RR, where RR is the risk ratio (proportion of subjects reporting events in the GSK257049 Comparator [6-12W] Group over the proportion in Menjugate Comparator [6-12W] Group); Test type: Superiority; p = 0.6280, Two-sided Fisher Exact test; Vaccine efficacy = -6.80, 95% CI 2-sided [-42.0 to 19.60]

7. Secondary Outcome: Number of Subjects With Prevalent Severe Anemia (Level of Hemoglobin <5g/dL)
Description: Prevalent severe anemia (PSA) was defined as a documented hemoglobin lower than (<) 5.0 grams per deciliter (g/dL), identified at an annual visit.
Time Frame: At Years 1, 2 and 3
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 [5-17M] Group | GSK257049 Comparator [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 [6-12W] Group | GSK257049 Comparator [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 565 | 528 | 562 | 437 | 436 | 421
Participants
  Prevalent severe anemia, Year 1: number analyzed (Participants) | 152 | 139 | 154 | 168 | 176 | 169
  Prevalent severe anemia, Year 1 | 0 | 0 | 0 | 0 | 0 | 0
  Prevalent severe anemia, Year 2 | 0 | 0 | 1 | 0 | 1 | 0
  Prevalent severe anemia, Year 3: number analyzed (Participants) | 561 | 516 | 550 | 434 | 408 | 411
  Prevalent severe anemia, Year 3 | 0 | 0 | 0 | 0 | 1 | 0
Statistical Analysis 1: Comparison: GSK257049 [5-17M] Group vs VeroRab Comparator [5-17M] Group; Vaccine efficacy (VE) against prevalent severe anemia assessed at Year 2 was estimated as 1-RR, where RR is the risk ratio (proportion of subjects reporting events in the GSK257049 [5-17M] Group over the proportion in VeroRab Comparator [5-17M] Group); Test type: Superiority; p = 0.4987, Two-sided Fisher Exact test; Vaccine efficacy = 100.0, 95% CI 2-sided [-3779 to 100.0]
Statistical Analysis 2: Comparison: GSK257049 Comparator [5-17M] Group vs VeroRab Comparator [5-17M] Group; Vaccine efficacy (VE) against prevalent severe anemia assessed at Year 2 was estimated as 1-RR, where RR is the risk ratio (proportion of subjects reporting events in the GSK257049 Comparator [5-17M] Group over the proportion in VeroRab Comparator [5-17M] Group); Test type: Superiority; p = 1.0000, Two-sided Fisher Exact test; Vaccine efficacy = 100.00, 95% CI 2-sided [-4051 to 100.0]

8. Secondary Outcome: Number of Subjects With Prevalent Moderate Anemia (Level of Hemoglobin <8g/dL)
Description: Prevalent moderate anemia (PMA) was defined as a documented hemoglobin < 8.0 g/dL, identified at an annual visit.
Time Frame: At Years 1, 2 and 3
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 [5-17M] Group | GSK257049 Comparator [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 [6-12W] Group | GSK257049 Comparator [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 565 | 528 | 562 | 437 | 436 | 421
Participants
  Prevalent moderate anemia, Year 1: number analyzed (Participants) | 152 | 139 | 154 | 168 | 176 | 169
  Prevalent moderate anemia, Year 1 | 7 | 9 | 2 | 16 | 6 | 11
  Prevalent moderate anemia, Year 2 | 7 | 10 | 11 | 18 | 15 | 8
  Prevalent moderate anemia, Year 3: number analyzed (Participants) | 561 | 516 | 550 | 434 | 408 | 411
  Prevalent moderate anemia, Year 3 | 4 | 4 | 7 | 10 | 6 | 8
Statistical Analysis 1: Comparison: GSK257049 [5-17M] Group vs VeroRab Comparator [5-17M] Group; Vaccine efficacy (VE) against prevalent moderate anemia assessed at Year 1 was estimated as 1-RR, where RR is the risk ratio (proportion of subjects reporting events in the GSK257049 [5-17M] Group over the proportion in VeroRab Comparator [5-17M] Group); Test type: Superiority; p = 0.1025, Two-sided Fisher Exact test; Vaccine efficacy = -254.60, 95% CI 2-sided [-3399 to 32.50]
Statistical Analysis 2: Comparison: GSK257049 Comparator [5-17M] Group vs VeroRab Comparator [5-17M] Group; Vaccine efficacy (VE) against prevalent moderate anemia assessed at Year 1 was estimated as 1-RR, where RR is the risk ratio (proportion of subjects reporting events in the GSK257049 Comparator [5-17M] Group over the proportion in VeroRab Comparator [5-17M] Group); Test type: Superiority; p = 0.0284, Two-sided Fisher Exact test; Vaccine efficacy = -398.60, 95% CI 2-sided [-4642 to -3.20]
Statistical Analysis 3: Comparison: GSK257049 [5-17M] Group vs VeroRab Comparator [5-17M] Group; Vaccine efficacy (VE) against prevalent moderate anemia assessed at Year 2 was estimated as 1-RR, where RR is the risk ratio (proportion of subjects reporting events in the GSK257049 [5-17M] Group over the proportion in VeroRab Comparator [5-17M] Group); Test type: Superiority; p = 0.3543, Two-sided Fisher Exact test; Vaccine efficacy = 36.70, 95% CI 2-sided [-78.8 to 79.20]
Statistical Analysis 4: Comparison: GSK257049 Comparator [5-17M] Group vs VeroRab Comparator [5-17M] Group; Vaccine efficacy (VE) against prevalent moderate anemia assessed at Year 2 was estimated as 1-RR, where RR is the risk ratio (proportion of subjects reporting events in the GSK257049 Comparator [5-17M] Group over the proportion in VeroRab Comparator [5-17M] Group); Test type: Superiority; p = 1.0000, Two-sided Fisher Exact test; Vaccine efficacy = 3.20, 95% CI 2-sided [-151 to 63.20]
Statistical Analysis 5: Comparison: GSK257049 [5-17M] Group vs VeroRab Comparator [5-17M] Group; Vaccine efficacy (VE) against prevalent moderate anemia assessed at Year 3 was estimated as 1-RR, where RR is the risk ratio (proportion of subjects reporting events in the GSK257049 [5-17M] Group over the proportion in VeroRab Comparator [5-17M] Group); Test type: Superiority; p = 0.3809, Two-sided Fisher Exact test; Vaccine efficacy = 44.00, 95% CI 2-sided [-120 to 88.00]
Statistical Analysis 6: Comparison: GSK257049 Comparator [5-17M] Group vs VeroRab Comparator [5-17M] Group; Vaccine efficacy (VE) against prevalent moderate anemia assessed at Year 3 was estimated as 1-RR, where RR is the risk ratio (proportion of subjects reporting events in the GSK257049 Comparator [5-17M] Group over the proportion in VeroRab Comparator [5-17M] Group); Test type: Superiority; p = 0.5490, Two-sided Fisher Exact test; Vaccine efficacy = 39.10, 95% CI 2-sided [-140 to 86.90]
Statistical Analysis 7: Comparison: GSK257049 [6-12W] Group vs Menjugate Comparator [6-12W] Group; Vaccine efficacy (VE) against prevalent moderate anemia assessed at Year 1 was estimated as 1-RR, where RR is the risk ratio (proportion of subjects reporting events in the GSK257049 [6-12W] Group over the proportion in Menjugate Comparator [6-12W] Group); Test type: Superiority; p = 0.3239, Two-sided Fisher Exact test; Vaccine efficacy = -46.30, 95% CI 2-sided [-249 to 36.20]
Statistical Analysis 8: Comparison: GSK257049 Comparator [6-12W] Group vs Menjugate Comparator [6-12W] Group; Vaccine efficacy (VE) against prevalent moderate anemia assessed at Year 1 was estimated as 1-RR, where RR is the risk ratio (proportion of subjects reporting events in the GSK257049 Comparator [6-12W] Group over the proportion in Menjugate Comparator [6-12W] Group); Test type: Superiority; p = 0.2184, Two-sided Fisher Exact test; Vaccine efficacy = 47.60, 95% CI 2-sided [-54.5 to 84.10]
Statistical Analysis 9: Comparison: GSK257049 [6-12W] Group vs Menjugate Comparator [6-12W] Group; Vaccine efficacy (VE) against prevalent moderate anemia assessed at Year 2 was estimated as 1-RR, where RR is the risk ratio (proportion of subjects reporting events in the GSK257049 [6-12W] Group over the proportion in Menjugate Comparator [6-12W] Group); Test type: Superiority; p = 0.0724, Two-sided Fisher Exact test; Vaccine efficacy = -116.80, 95% CI 2-sided [-476 to 10.30]
Statistical Analysis 10: Comparison: GSK257049 Comparator [6-12W] Group vs Menjugate Comparator [6-12W] Group; Vaccine efficacy (VE) against prevalent moderate anemia assessed at Year 2 was estimated as 1-RR, where RR is the risk ratio (proportion of subjects reporting events in the GSK257049 Comparator [6-12W] Group over the proportion in Menjugate Comparator [6-12W] Group); Test type: Superiority; p = 0.2055, Two-sided Fisher Exact test; Vaccine efficacy = -81.00, 95% CI 2-sided [-393 to 27.90]
Statistical Analysis 11: Comparison: GSK257049 [6-12W] Group vs Menjugate Comparator [6-12W] Group; Vaccine efficacy (VE) against prevalent moderate anemia assessed at Year 3 was estimated as 1-RR, where RR is the risk ratio (proportion of subjects reporting events in the GSK257049 [6-12W] Group over the proportion in Menjugate Comparator [6-12W] Group); Test type: Superiority; p = 0.8138, Two-sided Fisher Exact test; Vaccine efficacy = -18.40, 95% CI 2-sided [-245 to 57.90]
Statistical Analysis 12: Comparison: GSK257049 Comparator [6-12W] Group vs Menjugate Comparator [6-12W] Group; Vaccine efficacy (VE) against prevalent moderate anemia assessed at Year 3 was estimated as 1-RR, where RR is the risk ratio (proportion of subjects reporting events in the GSK257049 Comparator [6-12W] Group over the proportion in Menjugate Comparator [6-12W] Group); Test type: Superiority; p = 0.7887, Two-sided Fisher Exact test; Vaccine efficacy = 24.40, 95% CI 2-sided [-148 to 78.40]

9. Secondary Outcome: Incidence of Severe Malaria Meeting Case Definition 1.
Description: as for outcome 1
Time Frame: From Month 0 (study start of Malaria-055) to Year 3 (study end of Malaria-076)
Population: The analysis was performed on the modified Intention-to-Treat (ITT) population, which included all subjects that consented to the trial and received Dose 1 of the corresponding vaccine in Malaria-055 (NCT00866619) study. The analyses on the modified ITT population were performed per treatment assignment on subjects from both studies.
Measure: Number; unit: events per person-year
Arm/Group | GSK257049 [5-17M] Group | GSK257049 Comparator [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 [6-12W] Group | GSK257049 Comparator [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 844 | 829 | 839 | 637 | 635 | 633
events per person-year | 0.009 | 0.016 | 0.015 | 0.014 | 0.013 | 0.02
Statistical Analysis 1: Comparison: GSK257049 [5-17M] Group vs VeroRab Comparator [5-17M] Group; Vaccine efficacy (VE)/incidence comparison against all episodes of severe malaria were estimated as 1-incidence ratio (IR; total number of events/follow-up time in the GSK257049 [5-17M] Group over the total number of events/follow-up time in the VeroRab Comparator [5-17M] Group); Test type: Superiority; p = 0.0077, Negative binomial regression; Mixed model without random effect [Lievens, 2011]; Vaccine efficacy = 40.50, 95% CI 2-sided [12.84 to 59.39]
Statistical Analysis 2: Comparison: GSK257049 Comparator [5-17M] Group vs VeroRab Comparator [5-17M] Group; Vaccine efficacy (VE)/incidence comparison against all episodes of severe malaria were estimated as 1-incidence ratio (IR; total number of events/follow-up time in the GSK257049 Comparator [5-17M] Group over the total number of events/follow-up time in the VeroRab Comparator [5-17M] Group); Test type: Superiority; p = 0.7922, Negative binomial regression; Mixed model without random effect [Lievens, 2011]; Vaccine efficacy = -4.52, 95% CI 2-sided [-45.3 to 24.80]
Statistical Analysis 3: Comparison: GSK257049 [6-12W] Group vs Menjugate Comparator [6-12W] Group; Vaccine efficacy (VE)/incidence comparison against all episodes of severe malaria were estimated as 1-incidence ratio (IR; total number of events/follow-up time in the GSK257049 [6-12W] Group over the total number of events/follow-up time in the Menjugate Comparator [6-12W] Group); Test type: Superiority; p = 0.0802, Negative binomial regression; Mixed model without random effect [Lievens, 2011]; Vaccine efficacy = 29.03, 95% CI 2-sided [-4.22 to 51.67]
Statistical Analysis 4: Comparison: GSK257049 Comparator [6-12W] Group vs Menjugate Comparator [6-12W] Group; Vaccine efficacy (VE)/incidence comparison against all episodes of severe malaria were estimated as 1-incidence ratio (IR; total number of events/follow-up time in the GSK257049 Comparator [6-12W] Group over the total number of events/follow-up time in the Menjugate Comparator [6-12W] Group); Test type: Superiority; p = 0.0387, Negative binomial regression; Mixed model without random effect [Lievens, 2011]; Vaccine efficacy = 33.87, 95% CI 2-sided [2.13 to 55.32]

10. Secondary Outcome: Incidence of Severe Malaria Meeting Case Definition 2.
Description: as for outcome 2
Time Frame: From Month 0 (study start of Malaria-055) to Year 3 (study end of Malaria-076)
Population: as for outcome 9
Measure: Number; unit: events per person-year
Arm/Group | GSK257049 [5-17M] Group | GSK257049 Comparator [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 [6-12W] Group | GSK257049 Comparator [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 844 | 829 | 839 | 637 | 635 | 633
events per person-year | 0.015 | 0.021 | 0.023 | 0.019 | 0.019 | 0.028
Statistical Analysis 1: Comparison: GSK257049 [5-17M] Group vs VeroRab Comparator [5-17M] Group; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.0028, Negative binomial regression; Mixed model without random effect [Lievens, 2011]; Vaccine efficacy = 36.69, 95% CI 2-sided [14.60 to 53.07]
Statistical Analysis 2: Comparison: GSK257049 Comparator [5-17M] Group vs VeroRab Comparator [5-17M] Group; [analysis description as in outcome 9, analysis 2]; Test type: Superiority; p = 0.4430, Negative binomial regression; Mixed model without random effect [Lievens, 2011]; Vaccine efficacy = 10.14, 95% CI 2-sided [-18.1 to 31.64]
Statistical Analysis 3: Comparison: GSK257049 [6-12W] Group vs Menjugate Comparator [6-12W] Group; [analysis description as in outcome 9, analysis 3]; Test type: Superiority; p = 0.0245, Negative binomial regression; Mixed model without random effect [Lievens, 2011]; Vaccine efficacy = 30.99, 95% CI 2-sided [4.67 to 50.04]
Statistical Analysis 4: Comparison: GSK257049 Comparator [6-12W] Group vs Menjugate Comparator [6-12W] Group; [analysis description as in outcome 9, analysis 4]; Test type: Superiority; p = 0.0122, Negative binomial regression; Mixed model without random effect [Lievens, 2011]; Vaccine efficacy = 34.24, 95% CI 2-sided [8.74 to 52.61]

11. Secondary Outcome: Incidence of Clinical Malaria Meeting Case Definition
Description: Clinical malaria was defined as an episode of malaria with positive Plasmodium falciparum asexual parasitemia, accompanied by the presence of fever (axillary temperature ≥ 37.5°C) at the time of presentation or history of fever within 24 hours of presentation and occurring in a child who was unwell and brought for treatment to a healthcare facility. The incidence of clinical malaria for case definition 1 is expressed as a person year rate for each group (n/T), representing the number of events (n) reported over the risk period, which was counted in days and expressed as person years at risk (T). Due to late protocol approvals and retrospective data collection the sites did not collect the data according to protocol and as such the case definition cannot be applied. For the final analysis, specific case definitions based on available data were developed.
Time Frame: From Month 0 (study start of Malaria-055) to Year 3 (study end of Malaria-076)
Population: as for outcome 9
Measure: Number; unit: events per subject-year
Arm/Group | GSK257049 [5-17M] Group | GSK257049 Comparator [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 [6-12W] Group | GSK257049 Comparator [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 844 | 829 | 839 | 637 | 635 | 633
events per subject-year | 1.277 | 1.348 | 1.555 | 1.662 | 1.723 | 1.921
Statistical Analysis 1: Comparison: GSK257049 [5-17M] Group vs VeroRab Comparator [5-17M] Group; Vaccine efficacy (VE)/incidence comparison against all episodes of clinical malaria were estimated as 1-incidence ratio (IR; total number of events/follow-up time in the GSK257049 [5-17M] Group over the total number of events/follow-up time in the VeroRab Comparator [5-17M] Group); Test type: Superiority; p < .0001, Negative binomial regression; Mixed model with over-dispersion parameter estimated from the random effect [Lievens, 2011]; Vaccine efficacy = 23.67, 95% CI 2-sided [15.93 to 30.71]
Statistical Analysis 2: Comparison: GSK257049 Comparator [5-17M] Group vs VeroRab Comparator [5-17M] Group; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p < .0001, Negative binomial regression; Mixed model with over-dispersion parameter estimated from the random effect [Lievens, 2011]; Vaccine efficacy = 19.15, 95% CI 2-sided [10.81 to 26.71]
Statistical Analysis 3: Comparison: GSK257049 [6-12W] Group vs Menjugate Comparator [6-12W] Group; Vaccine efficacy (VE)/incidence comparison against all episodes of clinical malaria were estimated as 1-incidence ratio (IR; total number of events/follow-up time in the GSK257049 [6-12W] Group over the total number of events/follow-up time in the Menjugate Comparator [6-12W] Group); Test type: Superiority; p = 0.0009, Negative binomial regression; Mixed model with over-dispersion parameter estimated from the random effect [Lievens, 2011]; Vaccine efficacy = 15.55, 95% CI 2-sided [6.72 to 23.54]
Statistical Analysis 4: Comparison: GSK257049 Comparator [6-12W] Group vs Menjugate Comparator [6-12W] Group; Vaccine efficacy (VE)/incidence comparison against all episodes of clinical malaria were estimated as 1-incidence ratio (IR; total number of events/follow-up time in the GSK257049 Comparator [6-12W] Group over the total number of events/follow-up time in the Menjugate Comparator [6-12W] Group); Test type: Superiority; p = 0.0056, Negative binomial regression; Mixed model with over-dispersion parameter estimated from the random effect [Lievens, 2011]; Vaccine efficacy = 13.15, 95% CI 2-sided [4.05 to 21.39]

12. Secondary Outcome: Number of Subjects With Malaria Hospitalization Meeting Case Definition 1.
Description: as for outcome 4
Time Frame: From Month 0 (study start of Malaria-055) to Year 3 (study end of Malaria-076)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 [5-17M] Group | GSK257049 Comparator [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 [6-12W] Group | GSK257049 Comparator [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 844 | 829 | 839 | 637 | 635 | 633
Participants | 61 | 82 | 94 | 52 | 60 | 73
Statistical Analysis 1: Comparison: GSK257049 [5-17M] Group vs VeroRab Comparator [5-17M] Group; Vaccine efficacy (VE) was estimated as 1-the risk ratio (RR; proportion of subjects reporting events in the GSK257049 [5-17M] Group over the proportion in VeroRab Comparator [5-17M] Group), from Month 0 (study start of Malaria-055) to Year 3 (study end of Malaria-076); Test type: Superiority; p = 0.0053, Two-sided Fisher Exact test; Vaccine efficacy = 35.50, 95% CI 2-sided [10.00 to 54.00]
Statistical Analysis 2: Comparison: GSK257049 Comparator [5-17M] Group vs VeroRab Comparator [5-17M] Group; Vaccine efficacy (VE) was estimated as 1-the risk ratio (RR; proportion of subjects reporting events in the GSK257049 Comparator [5-17M] Group over the proportion in VeroRab Comparator [5-17M] Group), Month 0 (study start of Malaria-055) to Year 3 (study end of Malaria-076); Test type: Superiority; p = 0.4255, Two-sided Fisher Exact test; Vaccine efficacy = 11.70, 95% CI 2-sided [-20.0 to 35.20]
Statistical Analysis 3: Comparison: GSK257049 [6-12W] Group vs Menjugate Comparator [6-12W] Group; Vaccine efficacy (VE) was estimated as 1-the risk ratio (RR; proportion of subjects reporting events in the GSK257049 [6-12W] Group over the proportion in Menjugate Comparator [6-12W] Group), from Month 0 (study start of Malaria-055) to Year 3 (study end of Malaria-076); Test type: Superiority; p = 0.0479, Two-sided Fisher Exact test; Vaccine efficacy = 29.20, 95% CI 2-sided [-2.40 to 51.40]
Statistical Analysis 4: Comparison: GSK257049 Comparator [6-12W] Group vs Menjugate Comparator [6-12W] Group; Vaccine efficacy (VE) was estimated as 1-the risk ratio (RR; proportion of subjects reporting events in the GSK257049 Comparator [6-12W] Group over the proportion in Menjugate Comparator [6-12W] Group), from Month 0 (study start of Malaria-055) to Year 3 (study end of Malaria-076); Test type: Superiority; p = 0.2346, Two-sided Fisher Exact test; Vaccine efficacy = 18.10, 95% CI 2-sided [-16.9 to 42.80]

13. Secondary Outcome: Number of Subjects With Malaria Hospitalization Meeting Case Definition 2.
Description: as for outcome 5
Time Frame: From Month 0 (study start of Malaria-055) to Year 3 (study end of Malaria-076).
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 [5-17M] Group | GSK257049 Comparator [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 [6-12W] Group | GSK257049 Comparator [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 844 | 829 | 839 | 637 | 635 | 633
Participants | 60 | 79 | 93 | 54 | 60 | 75
Statistical Analysis 1: Comparison: GSK257049 [5-17M] Group vs VeroRab Comparator [5-17M] Group; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.0051, Two-sided Fisher Exact test; Vaccine efficacy = 35.90, 95% CI 2-sided [10.30 to 54.40]
Statistical Analysis 2: Comparison: GSK257049 Comparator [5-17M] Group vs VeroRab Comparator [5-17M] Group; Vaccine efficacy (VE) was estimated as 1-the risk ratio (RR; proportion of subjects reporting events in the GSK257049 Comparator [5-17M] Group over the proportion in VeroRab Comparator [5-17M] Group), from Month 0 (study start of Malaria-055) to Year 3 (study end of Malaria-076); Test type: Superiority; p = 0.3340, Two-sided Fisher Exact test; Vaccine efficacy = 14.00, 95% CI 2-sided [-17.3 to 37.10]
Statistical Analysis 3: Comparison: GSK257049 [6-12W] Group vs Menjugate Comparator [6-12W] Group; Vaccine efficacy (VE) was estimated as 1-the risk ratio (RR; proportion of subjects reporting events in the GSK257049 [6-12W] Group over the proportion in Meenjugate Comparator [6-12W] Group), from Month 0 (study start of Malaria-055) to Year 3 (study end of Malaria-076); Test type: Superiority; p = 0.0511, Two-sided Fisher Exact test; Vaccine efficacy = 28.50, 95% CI 2-sided [-2.90 to 50.50]
Statistical Analysis 4: Comparison: GSK257049 Comparator [6-12W] Group vs Menjugate Comparator [6-12W] Group; Vaccine efficacy (VE) was estimated as 1-the risk ratio (RR; proportion of subjects reporting events in the GSK257049 Comparator [6-12W] Group over the proportion in Meenjugate Comparator [6-12W] Group), from Month 0 (study start of Malaria-055) to Year 3 (study end of Malaria-076); Test type: Superiority; p = 0.1729, Two-sided Fisher Exact test; Vaccine efficacy = 20.30, 95% CI 2-sided [-13.5 to 44.20]

14. Secondary Outcome: Number of Subjects With Cerebral Malaria Meeting Both Case Definitions.
Description: Cerebral malaria was defined as a positive P. falciparum asexual parasitemia (within -1 to +3 days of admission), accompanied either by the presence of a marker of disease severity (a Blantyre score ≤ 2) or a SAE report with 'cerebral malaria' as preferred term.
Time Frame: From Year 0 to Year 3 (Starting January 2014 and ending December 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 [5-17M] Group | GSK257049 Comparator [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 [6-12W] Group | GSK257049 Comparator [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 594 | 561 | 593 | 459 | 456 | 442
Participants | 0 | 2 | 0 | 1 | 0 | 0

15. Secondary Outcome: Number of Subjects With Fatal Malaria Meeting Case Definition 1.
Description: Fatal malaria, case definition 1, was defined as a SAE report with preferred terms 'malaria', 'plasmodium falciparum infection', 'cerebral malaria' with confirmed positive Plasmodium falciparum asexual parasitemia associated with a fatal outcome (excludes planned admissions for medical investigation/care or elective surgery and trauma).
Time Frame: From Year 0 to Year 3 (Starting January 2014 and ending December 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 [5-17M] Group | GSK257049 Comparator [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 [6-12W] Group | GSK257049 Comparator [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 594 | 561 | 593 | 459 | 456 | 442
Participants | 1 | 2 | 0 | 0 | 0 | 0

16. Secondary Outcome: Number of Subjects With Fatal Malaria Meeting Case Definition 2.
Description: Fatal malaria, case definition 2, was defined as a SAE report with preferred terms 'malaria', 'plasmodium falciparum infection', 'cerebral malaria' associated with a fatal outcome.
Time Frame: From Year 0 to Year 3 (Starting January 2014 and ending December 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 [5-17M] Group | GSK257049 Comparator [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 [6-12W] Group | GSK257049 Comparator [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 594 | 561 | 593 | 459 | 456 | 442
Participants | 1 | 2 | 2 | 3 | 1 | 1
Statistical Analysis 1: Comparison: GSK257049 [5-17M] Group vs VeroRab Comparator [5-17M] Group; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.6244, Two-sided Fisher Exact test; Vaccine efficacy = 50.10, 95% CI 2-sided [-859 to 99.20]
Statistical Analysis 2: Comparison: GSK257049 Comparator [5-17M] Group vs VeroRab Comparator [5-17M] Group; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p = 1.0000, Two-sided Fisher Exact test; Vaccine efficacy = -5.70, 95% CI 2-sided [-1358 to 92.30]
Statistical Analysis 3: Comparison: GSK257049 [6-12W] Group vs Menjugate Comparator [6-12W] Group; [analysis description as in outcome 4, analysis 3]; Test type: Superiority; p = 0.6244, Two-sided Fisher Exact test; Vaccine efficacy = -188.90, 95% CI 2-sided [-15000 to 76.80]
Statistical Analysis 4: Comparison: GSK257049 Comparator [6-12W] Group vs Menjugate Comparator [6-12W] Group; [analysis description as in outcome 4, analysis 4]; Test type: Superiority; p = 1.0000, Two-sided Fisher Exact test; Vaccine efficacy = 3.10, 95% CI 2-sided [-7509 to 98.80]

17. Secondary Outcome: Number of Subjects With Cerebral Malaria
Description: as for outcome 14
Time Frame: From Month 0 (study start of Malaria-055) to Year 3 (study end of Malaria-076).
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 [5-17M] Group | GSK257049 Comparator [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 [6-12W] Group | GSK257049 Comparator [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 844 | 829 | 839 | 637 | 635 | 633
Participants | 4 | 10 | 2 | 3 | 2 | 0
Statistical Analysis 1: Comparison: GSK257049 [5-17M] Group vs VeroRab Comparator [5-17M] Group; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.6869, Two-sided Fisher Exact test; Vaccine efficacy = -98.80, 95% CI 2-sided [-2098 to 71.50]
Statistical Analysis 2: Comparison: GSK257049 Comparator [5-17M] Group vs VeroRab Comparator [5-17M] Group; [analysis description as in outcome 13, analysis 2]; Test type: Superiority; p = 0.0213, Two-sided Fisher Exact test; Vaccine efficacy = -406.00, 95% CI 2-sided [-4650 to -7.80]

18. Secondary Outcome: Number of Subjects With Fatal Malaria Meeting Case Definition 1.
Description: as for outcome 15
Time Frame: From Month 0 (study start of Malaria-055) to Year 3 (study end of Malaria-076).
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 [5-17M] Group | GSK257049 Comparator [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 [6-12W] Group | GSK257049 Comparator [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 844 | 829 | 839 | 637 | 635 | 633
Participants | 2 | 4 | 1 | 1 | 2 | 0
Statistical Analysis 1: Comparison: GSK257049 [5-17M] Group vs VeroRab Comparator [5-17M] Group; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 1.0000, Two-sided Fisher Exact test; Vaccine efficacy = -98.80, 95% CI 2-sided [-12000 to 89.60]
Statistical Analysis 2: Comparison: GSK257049 Comparator [5-17M] Group vs VeroRab Comparator [5-17M] Group; [analysis description as in outcome 13, analysis 2]; Test type: Superiority; p = 0.2154, Two-sided Fisher Exact test; Vaccine efficacy = -304.80, 95% CI 2-sided [-20000 to 59.90]

19. Secondary Outcome: Number of Subjects With Fatal Malaria Meeting Case Definition 2.
Description: as for outcome 16
Time Frame: From Month 0 (study start of Malaria-055) to Year 3 (study end of Malaria-076).
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 [5-17M] Group | GSK257049 Comparator [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 [6-12W] Group | GSK257049 Comparator [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 844 | 829 | 839 | 637 | 635 | 633
Participants | 5 | 7 | 4 | 4 | 6 | 1
Statistical Analysis 1: Comparison: GSK257049 [5-17M] Group vs VeroRab Comparator [5-17M] Group; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 1.0000, Two-sided Fisher Exact test; Vaccine efficacy = -24.30, 95% CI 2-sided [-526 to 73.30]
Statistical Analysis 2: Comparison: GSK257049 Comparator [5-17M] Group vs VeroRab Comparator [5-17M] Group; [analysis description as in outcome 13, analysis 2]; Test type: Superiority; p = 0.3834, Two-sided Fisher Exact test; Vaccine efficacy = -77.10, 95% CI 2-sided [-725 to 55.00]
Statistical Analysis 3: Comparison: GSK257049 [6-12W] Group vs Menjugate Comparator [6-12W] Group; [analysis description as in outcome 12, analysis 3]; Test type: Superiority; p = 0.3740, Two-sided Fisher Exact test; Vaccine efficacy = -297.50, 95% CI 2-sided [-19000 to 60.70]
Statistical Analysis 4: Comparison: GSK257049 Comparator [6-12W] Group vs Menjugate Comparator [6-12W] Group; [analysis description as in outcome 12, analysis 4]; Test type: Superiority; p = 0.1240, Two-sided Fisher Exact test; Vaccine efficacy = -498.10, 95% CI 2-sided [-27000 to 27.40]

20. Secondary Outcome: Number of Subjects Reporting Any, Related, Malaria and Fatal Serious Adverse Events (SAEs)
Description: Malaria SAEs were defined as SAEs coded by MedDRA preferred term level as 'malaria', 'Plasmodium falciparum infection' or 'cerebral malaria". A serious adverse event was any untoward medical occurrence that: resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization or resulted in disability/incapacity. SAEs disclosed in this outcome are any SAEs , fatal SAEs, those that were related to vaccine administration in the primary study MALARIA-055 PRI (110021) and malaria hospitalization.
Time Frame: From Year 0 to Year 3 (Starting January 2014 and ending December 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 [5-17M] Group | GSK257049 Comparator [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 [6-12W] Group | GSK257049 Comparator [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 594 | 560 | 593 | 457 | 455 | 440
Participants
  Any SAE(s) | 20 | 25 | 27 | 19 | 18 | 25
  Related SAE(s) | 0 | 0 | 0 | 0 | 0 | 0
  Malaria SAE(s) | 19 | 20 | 24 | 17 | 16 | 24
  Fatal SAE(s) | 2 | 7 | 5 | 3 | 3 | 2

21. Secondary Outcome: Number of Subjects Reporting Any Potential Immune-mediated Disorders (pIMDs) SAEs
Description: Potential immune-mediated diseases (pIMDs) are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology. Regardless of it being considered an AE or an SAE, it should have been reported per the SAE reporting rules.
Time Frame: From Year 0 to Year 3 (Starting January 2014 and ending December 2016)
Population: The analysis was performed on the modified Intention-to-Treat (ITT) population, which included all subjects that consented to the trial and received Dose 1 of the corresponding vaccine in Malaria-055 (NCT00866619) study. The analyses on the modified ITT population were performed per treatment assignment.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 [5-17M] Group | GSK257049 Comparator [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 [6-12W] Group | GSK257049 Comparator [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 594 | 560 | 593 | 457 | 455 | 440
Participants | 0 | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: Number of Subjects With Meningitis SAEs
Description: For the further evaluation of the safety signal of meningitis all the cases occurring during the study were reported as SAE. Meningitis is defined as an SAE coded at lowest level terms code, coded by MedDRA preferred term level as: 'meningitis', 'meningitis haemophilus', 'meningitis meningococcal', 'meningitis salmonella', 'meningitis pneumococcal', 'meningitis staphylococcal', 'meningitis tuberculous', 'meningitis herpes', 'meningitis candida', 'meningitis enterococcal', 'meningitis enteroviral', 'meningitis neonatal', 'meningitis toxoplasmal', 'meningitis mumps', 'meningitis cryptococcal', 'meningitis histoplasma', 'meningitis trypanosomal', 'Neurosyphilis', 'meningitis leptospiral', 'meningitis listeria', 'meningitis in sarcoidosis' (code in preferred term 'cerebral sarcoidosis'), 'meningitis bacterial', 'meningitis viral', 'meningitis aseptic', 'meningitis fungal'.
Time Frame: From Year 0 to Year 3 (Starting January 2014 and ending December 2016)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK257049 [5-17M] Group | GSK257049 Comparator [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 [6-12W] Group | GSK257049 Comparator [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 594 | 560 | 593 | 457 | 455 | 440
Participants
  Meningitis meningococcal | 0 | 0 | 1 | 1 | 0 | 0
  Meningitis | 0 | 0 | 0 | 1 | 0 | 1
  Meningitis bacterial | 0 | 0 | 0 | 0 | 0 | 1

23. Secondary Outcome: Antibody Concentrations Against Against Plasmodium Falciparum Circumsporozoite (Anti-CS)
Description: Antibody concentrations were assessed by enzyme-linked immunosorbent assay (ELISA) and presented as geometric mean titers (GMTs). Seropositivity anti-CS antibody cut-off was 0.5 EU/mL for Malaria-055 time points and 1.9 EU/mL for Malaria-076 time points.
Time Frame: At screening, 1 month post Dose 3 (Month 3), 18 months post Dose 3 (Month 20), 1 month post Dose 4 (Month 21), 12 months post Dose 4 (Month 32) (of Malaria-055) and at Years 1, 2 and 3 (of Malaria-076)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | GSK257049 [5-17M] Group | GSK257049 Comparator [5-17M] Group | VeroRab Comparator [5-17M] Group | GSK257049 [6-12W] Group | GSK257049 Comparator [6-12W] Group | Menjugate Comparator [6-12W] Group
Number analyzed (Participants) | 154 | 152 | 160 | 141 | 153 | 129
EU/mL
  At Month 3 of Malaria-055 | 671.8 [601.1 to 750.7] | 599.3 [534.0 to 672.5] | 0.3 [0.2 to 0.3] | 152.9 [121.4 to 192.4] | 169.0 [135.9 to 210.0] | 0.3 [0.2 to 0.3]
  At Month 20 of Malaria-055: number analyzed (Participants) | 146 | 146 | 145 | 134 | 144 | 128
  At Month 20 of Malaria-055 | 38.0 [31.1 to 46.5] | 40.3 [33.8 to 48.2] | 0.3 [0.3 to 0.3] | 4.2 [3.2 to 5.6] | 5.5 [4.2 to 7.2] | 0.3 [0.3 to 0.3]
  At Month 21 of Malaria-055: number analyzed (Participants) | 143 | 146 | 146 | 131 | 145 | 126
  At Month 21 of Malaria-055 | 368.6 [329.1 to 412.9] | 38.8 [32.5 to 46.2] | 0.3 [0.3 to 0.3] | 149.3 [119.4 to 186.6] | 5.3 [4.0 to 6.9] | 0.3 [0.3 to 0.4]
  At Month 32 of Malaria-055: number analyzed (Participants) | 146 | 150 | 145 | 125 | 142 | 125
  At Month 32 of Malaria-055 | 54.7 [47.3 to 63.3] | 21.1 [17.6 to 25.2] | 0.3 [0.3 to 0.3] | 11.7 [8.6 to 16.0] | 3.6 [2.9 to 4.6] | 0.4 [0.3 to 0.4]
  At Year 1 of Malaria-076: number analyzed (Participants) | 51 | 47 | 46 | 45 | 56 | 49
  At Year 1 of Malaria-076 | 20.5 [15.3 to 27.5] | 13.6 [10.0 to 18.5] | 1.3 [1.0 to 1.5] | 5.9 [3.8 to 9.1] | 2.5 [1.9 to 3.2] | 1.4 [1.1 to 1.7]
  At Year 2 of Malaria-076: number analyzed (Participants) | 134 | 140 | 137 | 117 | 130 | 127
  At Year 2 of Malaria-076 | 14.9 [12.7 to 17.6] | 6.8 [5.7 to 8.2] | 1.2 [1.1 to 1.4] | 5.4 [4.2 to 6.8] | 2.4 [2.0 to 2.9] | 1.2 [1.1 to 1.3]
  At Year 3 of Malaria-076: number analyzed (Participants) | 132 | 134 | 130 | 125 | 127 | 124
  At Year 3 of Malaria-076 | 11.2 [9.4 to 13.4] | 5.0 [4.2 to 6.0] | 1.2 [1.1 to 1.4] | 3.9 [3.1 to 4.9] | 2.2 [1.9 to 2.6] | 1.2 [1.1 to 1.4]

ADVERSE EVENTS:
Time Frame: Serious Adverse Events (SAEs): during the entire follow-up period, from Year 0 to Year 3 (Starting January 2014 and ending December 2016).
Description: Safety results include data for subjects who had a signed ICF for study Malaria-076 by the parent(s)/LAR(s), including SAE data from subjects who were not enrolled in study Malaria-076 but had a reason for non-participation (death) collected. Solicited and unsolicited AE(s) were not collected during this study.
Arm/Group | GSK257049 Group | GSK257049 Comparator Group | VeroRab/Menjugate Comparator Group
All-Cause Mortality (participants affected / at risk) | 5/1051 | 10/1015 | 7/1033
Serious Adverse Events (participants affected / at risk) | 39/1051 | 43/1015 | 52/1033
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK257049 Group (N=1051) | GSK257049 Comparator Group (N=1015) | VeroRab/Menjugate Comparator Group (N=1033)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 6 (6) | 10 (11)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sickle cell anaemia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal mass (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acute abdomen (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholera (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Malaria (Infections and infestations) | 36 (38) | 36 (36) | 48 (56)
Meningitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Meningitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Meningitis meningococcal (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Salmonellosis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Typhoid fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Hemiplegia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2015-04-15): https://cdn.clinicaltrials.gov/large-docs/16/NCT02207816/Prot_000.pdf
  • Statistical Analysis Plan (2015-10-12): https://cdn.clinicaltrials.gov/large-docs/16/NCT02207816/SAP_001.pdf